CLINICAL TRIAL: NCT05372029
Title: Enhancing Treatment Outcomes Among Veterans With Alcohol Use Disorder: Clinical and Neural Markers of Adjunctive Approach-avoidance Training
Brief Title: AAT for Alcohol Use Disorder in Veterans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D3793-R
Record Dates: First submitted 2022-05-09; First posted 2022-05-12 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Alcohol Use Disorder
Keywords: alcohol; cognitive training; intervention; neuroimaging
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: Two group randomized controlled trial of AAT versus comparator
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization will occur using a code corresponding to intervention arm. Participant and provider will not know the number-condition link.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Approach Avoidance Training (Experimental): AAT condition, participants use a joystick to respond to the color of the border surrounding the stimulus images presented (i.e., "pull for green, push for blue"). The stimuli used are alcohol-related images and neutral beverage images. To experimentally manipulate automatic action tendencies, a contingency is set between alcohol stimuli and avoidance behaviors
  Interventions: Behavioral: Approach Avoidance Training
- Sham Training (Sham Comparator): In the Sham participants use a joystick to respond to the color of the border surrounding stimulus images presented. There is no contingency between instruction type and pictures (i.e., non-training version of the task)
  Interventions: Behavioral: Sham Training

INTERVENTIONS:
Behavioral: Approach Avoidance Training — AAT condition, participants use a joystick to respond to the color of the border surrounding the stimulus images presented (i.e., "pull for green, push for blue"). The stimuli used are alcohol-related images and neutral beverage images. To experimentally manipulate automatic action tendencies, a contingency is set between alcohol stimuli and avoidance behaviors
  Other Names: AAT
  Arms: Approach Avoidance Training
Behavioral: Sham Training — In the Sham participants use a joystick to respond to the color of the border surrounding stimulus images presented. There is no contingency between instruction type and pictures (i.e., non-training version of the task)
  Arms: Sham Training

SUMMARY:
The proposed study will test a novel treatment for alcohol use disorders (AUD) to determine if it helps Veterans reduce their hazardous drinking and recover from alcohol-related functional impairments across social, occupational, and domestic domains. To do so, the investigators will evaluate clinical, cognitive, and neural effects of a computer-delivered Approach Avoidance Training (AAT) treatment - which changes implicit tendencies to approach alcohol-related cues - in conjunction with standard VA care. The project will support RR&D's mission to improve Veterans' participation in their lives and community by determining if this innovative alternative technique can improve recovery outcomes for Veterans with AUD and exploring how the intervention works.

DETAILED DESCRIPTION:
Veterans with alcohol use disorders (AUD) would be greatly served by development of effective interventions to address high relapse rates and difficulty with resuming optimal functional recovery (i.e., re-engaging in vocational, social, and daily life roles that are critical to maintaining alcohol consumption goals). Approach bias toward alcohol, an implicit motivational response to alcohol cues observable across behavioral and neural indicators, is a core feature of AUD that impedes recovery but is not routinely treated in standard care. Treatment options that target approach bias may improve outcomes by decreasing the appetitive pull of alcohol, so that individuals are better able to disengage from habitual drinking behaviors in the service of their functional goals and objectives. Approach Avoidance Training (AAT) is a computer-delivered treatment program that shifts behavioral and neural indicators of approach bias for alcohol and has been shown to improve drinking-related outcomes in AUD when used in conjunction with standard care. Given the promise of this intervention for AUD, there is a critical need to determine if this treatment can be successfully used for Veterans who commonly present with complex comorbidities, and to pinpoint cognitive and neurobiological processes of change. The overall objectives of this proposal are to determine whether Alcohol Approach Avoidance Training (AAT) improves recovery outcomes in Veterans undergoing standard care for AUD with co-occurring conditions, and to identify the underlying cognitive and neural substrates modified. The central hypothesis is that AAT training will improve critical recovery outcomes for Veterans and improve behavioral and neural indicators of approach bias. The investigators will explore whether effects of AAT generalize to related top-down and bottom-up neurocognitive processes. The investigators will also explore potential predictors of treatment response. The overall objectives will be addressed in a randomized controlled trial of 136 Veterans completing standard care in the local VA setting with either AAT or a control condition. Aim 1 will determine if repeatedly practicing avoidance of alcohol cues through AAT can improve recovery outcomes and hazardous drinking. Aim 2 will determine if AAT modifies approach bias by measuring this construct with multiple assessment methods (i.e., behavioral, fMRI). Exploratory aims will examine if AAT modifies inhibition (top-down) and cue reactivity (bottom up) processing, and the extent to which baseline comorbidity severity, treatment engagement characteristics, or baseline approach bias (behavioral task reaction times, brain response during fMRI) are associated with clinical outcomes. The project is expected to determine if AAT shows clinical potential that would warrant expansion to other substances of abuse and a larger multisite confirmatory efficacy trial in Veterans with AUD. Results of the study will inform the utility of AAT as an adjunctive AUD treatment for Veterans, potentially offering a novel, low-cost, and portable alternative option to improve recovery in these individuals. Consistent with the RR&D mission to maximize "functional independence, quality of life and participation in their lives and community," the project will provide a foundation for neuroscience-based alternative therapeutic options to improve recovery in Veterans with AUD.

ELIGIBILITY:
Inclusion Criteria:

* fluent in English
* primary diagnosis of AUD with no more than 90 days abstinence from alcohol
* 4-week stability if taking psychotropic medications

Exclusion Criteria:

* lifetime history of psychotic or bipolar disorder
* neurodegenerative or neurodevelopmental disorders
* history of moderate or severe traumatic brain injury or other known neurological condition
* sensory deficits that would preclude completing tasks
* suicidal or homicidal ideation within the past month necessitating urgent higher level care
* concurrent individual psychotherapy or other treatment outside of standard DDRP programming
* conditions unsafe for completing MRI scanning for those completing the scanning component only (e.g., metal in body)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in the Drinker Inventory of Consequences (DrInC) | Baseline, post (week 6), follow up 1 (3 mo.), followup 2 (6 mo.)
  The DrInC assesses alcohol-related adverse functional consequences across physical (e.g., harmed physical health), interpersonal (e.g., loss of relationships), role responsibilities (e.g., missed work), psychological (e.g., loss of hobbies), and impulse control-related problems (e.g., legal problems) with higher scores indicating worse outcomes. Total scores range from 0 to 50.

SECONDARY OUTCOMES:
Change in the Timeline Follow-back Procedure (TLFB) | Baseline, post (week 6), follow up 1 (3 mo.), followup 2 (6 mo.)
  The TLFB evaluates drinking and all drug use during the 90 days preceding interviews. Percent heavy drinking days ranges from 0-100% with higher indicating more days.
Change in Alcohol Approach Avoidance Behavioral Assessment (approach bias score) | Baseline, post (week 6)
  Participants must pull or push alcohol or neutral cues using a joystick. The outcome approach bias score is computed by subtracting each participant's mean response latency in the pull condition from his or her mean response latency in the corresponding push condition (e.g., alcohol-push minus alcohol-pull). Higher scores indicate higher approach bias.
Change in Alcohol Approach Avoidance Imaging Assessment (BOLD neural signal) | Baseline, post (week 6)
  Participants must pull or push alcohol or neutral cues using a joystick while undergoing functional MRI. The outcome is BOLD percent signal change to a contrast comparing alcohol to neutral beverage for push versus pull. Higher scores indicate higher percent signal change.

OTHER OUTCOMES:
Change in Sheehan Disability Scale (SDS) | Baseline, post (week 6), follow up 1 (3 mo.), followup 2 (6 mo.)
  The SDS assesses functional impairment due to clinical symptoms across three domains: work/school, social functioning, and family life. Higher scores indicate higher functional impairment. Domain scores range from 0-10.
Change in The Substance Use Recovery Evaluator (SURE) | Baseline, post (week 6), follow up 1 (3 mo.), followup 2 (6 mo.)
  The SURE measures alcohol recovery along the following domains: substance use, material resources, self-care, relationships, and outlook on life. Higher scores indicate worse recovery outcomes. Total scores range from 21-63.
Change in Alcohol Inhibition fMRI task (BOLD neural signal) | Baseline, post (week 6)
  Participants are shown an alcohol or neutral cue and must decide to respond or not respond as quickly as possible. The outcome is BOLD percent signal change to a contrast comparing inhibition versus non-inhibition trials. Higher scores indicate higher percent signal change.
Change in Alcohol Cue Reactivity fMRI task | Baseline, post (week 6)
  Participants passively view alcohol or neutral cues. The outcome is BOLD percent signal change to a contrast comparing alcohol cues to non-alcohol cue trials. Higher scores indicate higher percent signal change.
Stages of Change Readiness and Eagerness Scale (SOCRATES) | Baseline, post (week 6), follow up 1 (3 mo.), followup 2 (6 mo.)
  The SOCRATES measures readiness to change drinking related behavior with higher scores indicating greater readiness to change.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica A Bomyea, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Caudle MM, Klaming R, Fong C, Harle K, Taylor C, Spadoni A, Bomyea J. Approach avoidance training versus Sham in veterans with alcohol use disorder: protocol for a randomized controlled trial. BMC Psychiatry. 2023 Jul 12;23(1):499. doi: 10.1186/s12888-023-04961-z. PMID 37438722